CLINICAL TRIAL: NCT04763798
Title: Efficacy of Hamstring Stretching According to the Neural or Muscle Tissue Involvement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat Internacional de Catalunya (Other)
Responsible Party: Principal Investigator, Carlos López de Celis, Doctor, Universitat Internacional de Catalunya
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CBAS-2019-12
Record Dates: First submitted 2021-02-12; First posted 2021-02-21 (Actual); Last update posted 2022-09-06 (Actual); Status verified 2021-02

CONDITIONS: Muscle Stretching
Keywords: Hamstring; Passive Knee extension test; Straight-leg-raise; maximun hip flexion; musculoskeletal response; nerve response

STUDY DESIGN:
Intervention Model Description: Cross sectional study. Randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: A single-blind (evaluator) randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dominant (Experimental): All subjects will receive the three stretching techniques on dominant leg. Interventions will be performed in three different days and only one of the three stretching exercises will be performed in each session. The rest period between sessions will be one week. Stretching exercises will be perform in a random order. A random-number generator will be used for randomization
  Interventions: Other: Straight-leg-raise (SLR); Other: Passive Knee extension test (PKE); Other: Maximum hip flexion (MHF)
- Non dominant (Active Comparator): All subjects will receive the three stretching techniques on non dominant leg. Interventions will be performed in three different days and only one of the three stretching exercises will be performed in each session. The rest period between sessions will bé one week. Stretching exercises will be perform in a random order. A random-number generator will bé used for randomization
  Interventions: Other: Straight-leg-raise (SLR); Other: Passive Knee extension test (PKE); Other: Maximum hip flexion (MHF)

INTERVENTIONS:
Other: Straight-leg-raise (SLR) — The stretched lower limb was on a mobile support and the contralateral limb was stabilized with a belt on the bench. For the SLR, the knee was kept in full extension and then, hip flexion was performed until a marked resistance. All stretching modalities were applied until a marked resistance was felt by the physical therapist (end-feel) or until the point of maximal tolerance referred by subjects.The stretch lasted 30 seconds followed by 15 seconds rest period and the procedure was repeated 5 times. Each stretching was applied for 5 minutes
Other: Passive Knee extension test (PKE) — The stretched lower limb was on a mobile support and the contralateral limb was stabilized with a belt on the bench. For the PKE, the hip was kept in 90º flexion and then, knee extension was performed. All stretching modalities were applied until a marked resistance was felt by the physical therapist (end-feel) or until the point of maximal tolerance referred by subjects.
  The stretches lasted 30 seconds followed by 15 seconds rest period and the procedure was repeated 5 times. Each stretching was applied for 5 minutes
Other: Maximum hip flexion (MHF) — The stretched lower limb was on a mobile support and the contralateral limb was stabilized with a belt on the bench. For MHF, a maximal hip flexion was performed and then, knee extension was applied. All stretching modalities were applied until a marked resistance was felt by the physical therapist (end-feel) or until the point of maximal tolerance referred by subjects.
  The stretches lasted 30 seconds followed by 15 seconds rest period and the procedure was repeated 5 times. Each stretching was applied for 5 minutes

SUMMARY:
Background: Muscle stretching is a technique widely used in the clinical practice of physiotherapy and in the field of sports. In the bibliography we find a multitude of stretches and procedures described, some of them being similar to neurodynamic tests, which could direct their effect to a neural and not a musculoskeletal structure. The structural differentiation manoeuvre has been shown to be able to discriminate the increase in tension on the nerve.

Objective: To evaluate the short-term efficacy on ischiosural muscle elongation of three modalities of ischiosural stretching according to neural or muscular involvement, in subjects without previous pathology.

Design: Cross sectional study. Methods: A randomised, blinded, assessor-blinded clinical trial was performed. According to the sample size calculation, a total of 35 subjects will be recruited from the International University of Catalonia. Each subject will undergo three hamstring stretching techniques on their dominant leg, Straight-leg-raise (SLR), Passive knee extension (PKE) and Maximun hip flexion (MHF) with an interval of one week on the dominant leg. Muscle elongation in each stretching modality will be assessed with the modified black saver sit and reach test and whether the technique generates a neural or musculoskeletal response when performing the structural differentiation manoeuvre.

DETAILED DESCRIPTION:
Background: Muscle stretching is a technique widely used in the clinical practice of physiotherapy and in the field of sports. In the bibliography we find a multitude of stretches and procedures described, some of them being similar to neurodynamic tests, which could direct their effect to a neural and not a musculoskeletal structure. The structural differentiation manoeuvre has been shown to be able to discriminate the increase in tension on the nerve.

Objective: To evaluate the short-term efficacy on ischiosural muscle elongation of three modalities of ischiosural stretching according to neural or muscular involvement, in subjects without previous pathology.

Design: Cross sectional study.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects over 18 years old who signed the informed consent.

Exclusion Criteria:

* The exclusion criteria were as follows: 1) injury in the thigh 6 months previously, 2) diagnosis of any orthopaedic problem or surgery in the lower limbs, 3) back pain or previous surgery in the spine or 4) systemic or neurological disorders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2020-12-11 (Actual); Primary Completion 2021-01-11 (Actual); Study Completion 2021-02-20 (Actual)

PRIMARY OUTCOMES:
Modified back-saver sit-and-reach test | Through study completion, an average of 3 weeks.
  subjects will perform a single-leg sit-and-reach on a bench. The untested leg will be placed on the floor with knee at approximately 90º. A measuring tape will be placed on the bench. Subjects aligned the sole of the foot of the tested leg with the 50-cm mark on the measuring tape. Thereafter, subjects will be asked to reach forward as far as possible while maintaining the knees, arms, and fingers fully extended, and keep in the two hands on tip of each other and palms down
Distal sensation | Through study completion, an average of 3 weeks.
  Passive ankle dorsiflexion was performed as distal sensation manoeuvre at the final position of all stretching modalities. Subjects were asked to indicate if the sensation during the stretching was modified during the ankle dorsiflexion (neural response) or was the same (musculoskeletal response)
Force intensity applyed | Through study completion, an average of 3 weeks.
  The intensity of the force applied during each stretching modality was measured by a manual dynamometer (MicroFET2, Hoggan Scientific, Salt Lake City, Utah). The dynamometer was applied on the distal leg, proximal to the ankle joint. The physiotherapist performed the stretching until a marked resistance was felt and then, the force was registered.

SECONDARY OUTCOMES:
Perceived sensation | Through study completion, an average of 3 weeks.
  After the stretching application, all subjects were asked about their perceived sensation. They were asked about the intensity of the tension sensation during the technique. A numeric scale, ranging from 0 ("no tension") to 10 ("worst tension imaginable") was used to indicate the intensity of tension sensation during the stretching technique.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos L López de Celis, Dr, Principal Investigator — Universitat Internacional de Catalunya
Locations (1):
- Universitat Internacional de Catalunya, Sant Cugat del Vallès, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided